CLINICAL TRIAL: NCT02509403
Title: An Open-label Trial to Evaluate the Safety of an Essential Oil Infused Perineal Towel - WIPEAWAY
Brief Title: An Open-label Trial to Evaluate the Safety of an Essential Oil Infused Perineal Towel
Acronym: WIPEAWAY
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The company responsible for funding has filed for bankruptcy
Sponsor: University of Alberta (Other)
Collaborators: Taiga BioActives Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAI-WA-0707
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Urinary Tract Infections
Keywords: Perineal hygiene; Hygiene wipes; Hygiene Towels; Safety; Essential oils; Natural Health Product
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Essential oils infused Perineal Hygiene wipe
  Interventions: Drug: Essential oils infused Perineal Hygiene wipe

INTERVENTIONS:
Drug: Essential oils infused Perineal Hygiene wipe — Each participant will be asked to complete a treatment period of one month's duration. At the start of the study, the participants will be asked to fill-out a baseline questionnaire and will be given a month's supply of the perineal hygiene towel with instructions about its use. At day 15, 30 and 45 follow-ups will be conducted.

SUMMARY:
The purpose of this study is to assess the safety (absence of skin irritation) of a feminine hygiene product for perineal hygiene prior to undertaking a clinical effectiveness trial. The feminine hygiene towel or wipe is an anti-bacterial Natural Health Product solution.

DETAILED DESCRIPTION:
The design of the trial will be open-label and uncontrolled.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years willing to use the perineal towels for an entire month

Exclusion Criteria:

* Pregnancy or within 12 months post-partum
* Current vulvo-vaginitis
* Known allergies to tea-tree oil

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants without any adverse events as a measure of safety | 45 Days
  Number of participants without any adverse events

SECONDARY OUTCOMES:
Ease of use of the perineal hygiene wipe by the participants on a daily basis | 30 Days
  Ease of use of the perineal hygiene wipe by the participants on a daily basis
Self-reported comfort score on a scale of 1 to 10 | 30 Days
  Self-reported comfort score on a scale of 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Wagg, MD, Principal Investigator — University of Alberta
Locations (1):
- Division of Geriatric Medicine, Clinical Sciences Building, University of Alberta Hosp, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Foxman B. Epidemiology of urinary tract infections: incidence, morbidity, and economic costs. Am J Med. 2002 Jul 8;113 Suppl 1A:5S-13S. doi: 10.1016/s0002-9343(02)01054-9. PMID 12113866
- [Background] Dason S, Dason JT, Kapoor A. Guidelines for the diagnosis and management of recurrent urinary tract infection in women. Can Urol Assoc J. 2011 Oct;5(5):316-22. doi: 10.5489/cuaj.11214. No abstract available. PMID 22031610
- [Background] Persad S, Watermeyer S, Griffiths A, Cherian B, Evans J. Association between urinary tract infection and postmicturition wiping habit. Acta Obstet Gynecol Scand. 2006;85(11):1395-6. doi: 10.1080/00016340600936977. PMID 17091423
- [Background] Amiri FN, Rooshan MH, Ahmady MH, Soliamani MJ. Hygiene practices and sexual activity associated with urinary tract infection in pregnant women. East Mediterr Health J. 2009 Jan-Feb;15(1):104-10. PMID 19469432
- [Background] Temple JG. Perineal hygiene in the prevention of recurring cystitis in women. Proc R Soc Med. 1972 Feb;65(2):169. doi: 10.1177/003591577206500222. No abstract available. PMID 5085024
- [Background] Leydon GM, Turner S, Smith H, Little P; UTIS team. Women's views about management and cause of urinary tract infection: qualitative interview study. BMJ. 2010 Feb 5;340:c279. doi: 10.1136/bmj.c279. PMID 20139217